CLINICAL TRIAL: NCT01791751
Title: Impact of Clomiphene Citrate Administration During the Early Luteal Phase on Endocrine Profile in Agonist Triggered GnRH Antagonist in Vitro Fertilization Cycles. Phase IV, Single-centre, Open-label, Controlled Clinical Trial.
Brief Title: Impact of Clomiphene Citrate Administration During the Early Luteal Phase on Endocrine Profile in IVF Cycles
Acronym: CLOFA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Privada Eugin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CLOFA; 2011-002173-33 (EudraCT Number)
Record Dates: First submitted 2012-11-12; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clomifene Citrate (Experimental): Clomifene Citrate 50 mg
  Interventions: Drug: Clomifene Citrate
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Clomifene Citrate — Clomiphene citrate 100 mg daily for 5 days
  Arms: Clomifene Citrate

SUMMARY:
The purpose of this study is to evaluate the effect on LH levels of the 5-day CC administration during luteal phase in oocyte donors, to investigate whether the CC corrects the suppressed LH levels in the luteal phase and whether it prolongs the luteal phase in the agonist triggered antagonist cycles.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors
* 18-35 years old
* BMI 18-29 Kg/m2
* Normal basal hormonal levels
* No contraceptive pill

Exclusion Criteria:

* Polycystic ovarian syndrome (PCOS)
* Previous participation in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
LH Levels (IU) | Luteal phase (up to 2 weeks)

SECONDARY OUTCOMES:
Endometrial development (Noyes criteria) | Luteal phase (1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Colodron, MD, Principal Investigator — Clinica EUGIN
Locations (1):
- Clínica EUGIN, Barcelona, Barcelona, Spain